CLINICAL TRIAL: NCT01944631
Title: Efficacy and Safety of Iota-Carrageenan Nasal Spray 1.2 g/l (0.12 Percent) (Bisolviral) Versus Placebo Nasal Spray in the Early Treatment of Common Cold
Brief Title: Iota-Carrageenan Nasal Spray in Common Cold
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1326.1
Record Dates: First submitted 2013-09-13; First posted 2013-09-17 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

ARMS (2):
- Placebo (Placebo Comparator): Nasal spray 4 times a day over 4 to 10 days
  Interventions: Device: Placebo
- Iota-Carrageenan nasal spray (Experimental): Nasal spray 4 times a day over 4 to 10 days
  Interventions: Device: Iota-Carrageenan

INTERVENTIONS:
Device: Placebo — Nasal spray saline
  Arms: Placebo
Device: Iota-Carrageenan — Nasal spray containing 1.20 g/l Iota-Carrageenan in saline
  Arms: Iota-Carrageenan nasal spray

SUMMARY:
The aim of this clinical trial is to investigate the effect of Iota-Carrageenan treatment on cold symptoms. The effect of treatment on the duration of the cold and the patients viral load plus cytokine level indicating the inflammatory response will be analyzed.

ELIGIBILITY:
Inclusion criteria:

* Patients consider that they are in an early stage of common cold with symptoms of no more than 48 hours duration
* Symptom score of equal or more than 1 for for at least one of the symptoms sore throat, runny nose and blocked nose on a 0-3 verbal rating scale
* Total symptom score of equal or less 9 for symptoms headache, muscle ache, chilliness, sore throat, blocked nose, runny nose, cough, and sneezing measured on a 0-3 verbal rating scale
* Patients agree to refrain from taking any products intended to prevent, intervene in, or treat cough/colds/flu, starting at study entry and continuing through day 10 (e.g. those containing zinc, Echinacea); use of a daily multivitamin is allowed.

Exclusion criteria:

* Known hypersensitivity or are allergic to any component of the test device
* Clinically significant cardiovascular, endocrinological, neurological, respiratory, gastrointestinal disease or history or any current disease that is considered by the investigator as a reason for exclusion e.g. current allergic rhinitis, chronic obstructive pulmonary disease
* Severe nasal septum deviation or other condition that could cause nasal obstruction such as the presence of nasal polyps.
* History of nasal or sinus surgery that in the opinion of the investigator may influence symptom scores
* Taking any prescribed medication other than for contraception, that is considered by the investigator as a reason for exclusion e.g. systemic steroids, intranasal medicines, antibiotics
* Common cold or flu like symptoms for more than 48 hours.
* Recent (within the previous 2 days) intake of a common cold medicine that in the opinion of the investigator may influence symptom scores (analgesics, nasal decongestants, cough medicines)
* Current smoker (more than 10 cigarettes a day)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1326.1.44001 Boehringer Ingelheim Investigational Site, Cardiff, United Kingdom

REFERENCES:
- [Derived] Eccles R, Winther B, Johnston SL, Robinson P, Trampisch M, Koelsch S. Efficacy and safety of iota-carrageenan nasal spray versus placebo in early treatment of the common cold in adults: the ICICC trial. Respir Res. 2015 Oct 5;16:121. doi: 10.1186/s12931-015-0281-8. PMID 26438038

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients received an application of placebo nasal spray saline 4 times a day, for 4 to 10 days. One application means one puff into each nostril.
- Bisolviral: Patients received an application of 1.20g/l Iota-Carrageenan in saline nasal spray 4 times a day, for 4 to 10 days. One application means one puff into each nostril.
Period: Overall Study
Arm/Group | Placebo | Bisolviral
Started | 100 | 100
Completed | 96 | 98
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set which included all randomised patients who used at least one dose of trial treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bisolviral | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.93 (1.90) | 20.01 (2.37) | 19.97 (2.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 122
  Male | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Total Symptom Score (TSS) Over Days 2 to 4 (TSS2-4)
Description: The total symptom score (TSS) is the sum of the 8 single common cold symptom scores consisting of 3 systemic (headache, muscle ache and chilliness) and 5 local (sore throat, blocked nose, runny nose, cough and sneezing) symptoms.
  Each common cold symptom was scored on a 4-point ordinal scale:
  * 0 = symptom not present
  * 1 = mild symptom (I can feel it but it has not disturbed or irritated me)
  * 2 = moderate symptom (symptom has disturbed and irritated me some of the time)
  * 3 = severe symptom (symptom has disturbed and irritated me most of the time)
  The mean over days 2 to 4 (TSS2-4) was calculated as (TSS2 + TSS3 + TSS4)/3 where TSS2, TSS3 and TSS4 are the total symptom scores calculated for days 2, 3 and 4 respectively. TSS2-4 ranges from 0 (no symptoms) to 24 (severe symptoms).
Time Frame: Days 2, 3 and 4
Population: Full analysis set (FAS) which included all randomised patients who used at least one dose of trial treatment, who provided a baseline total symptom score (TSS) as well as any post-treatment data for the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Patient received an application of placebo nasal spray saline 4 times a day, for 4 to 10 days. One application means one puff into each nostril.
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
units on a scale | 6.390 (0.254) | 5.777 (0.253)
Statistical Analysis 1: Comparison: Placebo vs Bisolviral; Test type: Superiority or Other; p = 0.0895, ANCOVA; Mean Difference (Net) = -0.613, 95% CI 2-sided [-1.321 to 0.095], Standard Error of Mean 0.359 — Difference calculated as bisolviral minus placebo

2. Secondary Outcome: Mean of the Sum of 3 Single Systemic Common Cold Symptom Scores Over Days 2 to 4 (SSS2-4)
Description: The mean of the sum of 3 single systemic common cold symptom scores (headache, muscle ache, chilliness).
  Each common cold symptom was scored on a 4-point ordinal scale:
  * 0 = symptom not present
  * 1 = mild symptom (I can feel it but it has not disturbed or irritated me)
  * 2 = moderate symptom (symptom has disturbed and irritated me some of the time)
  * 3 = severe symptom (symptom has disturbed and irritated me most of the time)
  The mean of the sum of 3 single systemic common cold symptom scores over days 2-4 was calculated as (SSS2 + SSS3 + SSS4)/3 where SSS2, SSS3 and SSS4 are the systemic common cold symptom scores calculated for days 2, 3 and 4 respectively. SSS2-4 ranges from 0 (no symptoms) to 9 (severe symptoms).
Time Frame: Days 2, 3 and 4
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
units on a scale | 1.297 (0.103) | 1.121 (0.103)
Statistical Analysis 1: Comparison: Bisolviral; Test type: Superiority or Other; p = 0.2310, ANCOVA; Mean Difference (Net) = -0.176, 95% CI 2-sided [-0.464 to 0.113], Standard Error of Mean 0.146 — Difference calculated as bisolviral minus placebo

3. Secondary Outcome: Mean of the Sum of 5 Single Local Common Cold Symptom Scores Mean Over Days 2 to 4 (LSS2-4)
Description: The mean of the sum of 5 single local common cold symptom scores (sore throat, blocked nose, runny nose, cough and sneezing).
  Each common cold symptom was scored on a 4-point ordinal scale:
  * 0 = symptom not present
  * 1 = mild symptom (I can feel it but it has not disturbed or irritated me)
  * 2 = moderate symptom (symptom has disturbed and irritated me some of the time)
  * 3 = severe symptom (symptom has disturbed and irritated me most of the time)
  The mean of the sum of 5 single local common cold symptom scores over days 2 to 4 was calculated as (LSS2 + LSS3 + LSS4)/3 where LSS2, LSS3 and LSS4 are the local common cold symptom scores calculated for days 2, 3 and 4 respectively. LSS2-4 ranges from 0 (no symptoms) to 15 (severe symptoms).
Time Frame: Days 2, 3 and 4
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
units on a scale | 5.100 (0.215) | 4.657 (0.214)
Statistical Analysis 1: Comparison: Placebo vs Bisolviral; Test type: Superiority or Other; p = 0.1465, ANCOVA; Mean Difference (Net) = -0.443, 95% CI 2-sided [-1.042 to 0.156], Standard Error of Mean 0.304 — Difference calculated as bisolviral minus placebo

4. Secondary Outcome: Area Under the Curve (AUC) Over the 10-day Period for the TSS (AUC-TSS 1-10)
Description: The total symptom score (TSS) is the sum of the 8 single common cold symptom scores consisting of 3 systemic (headache, muscle ache and chilliness) and 5 local (sore throat, blocked nose, runny nose, cough and sneezing) symptoms.
  Each common cold symptom was scored on a 4-point ordinal scale:
  * 0 = symptom not present
  * 1 = mild symptom (I can feel it but it has not disturbed or irritated me)
  * 2 = moderate symptom (symptom has disturbed and irritated me some of the time)
  * 3 = severe symptom (symptom has disturbed and irritated me most of the time)
  The Area under the curve (AUC) over the 10-day period for the total symptom score (AUC-TSS 1-10) was calculated as the sum of the TSS calculated on each day from day 1 to day 10. AUC-TSS 1-10 ranges from 0 (no symptoms) to 270 (severe symptoms).
Time Frame: Days 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale * days
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
units on a scale * days | 41.214 (2.199) | 41.941 (2.187)
Statistical Analysis 1: Comparison: Placebo vs Bisolviral; Test type: Superiority or Other; p = 0.8148, ANCOVA; Mean Difference (Net) = 0.728, 95% CI 2-sided [-5.390 to 6.845], Standard Error of Mean 3.102 — Difference calculated as bisolviral minus placebo

5. Secondary Outcome: Duration of the Cold
Description: Duration of the common cold was assessed by the question "Do you still have a cold?" at the end of each treatment day. The duration of the cold was defined as ended by the first day of a "No" answer to this daily question.
Time Frame: Baseline up to 10 days
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
days | 7 [7 to 8] | 8 [7 to 9]
Statistical Analysis 1: Comparison: Placebo vs Bisolviral; Test type: Superiority or Other; p = 0.1887, Log Rank; Log-rank test stratifying for the variable 'baseline TSS'

6. Secondary Outcome: Patient Overall Assessment of Efficacy
Description: Patient overall assessment of efficacy was assessed by the question "How effective was the treatment in relieving your common cold symptoms?" at day 10. A 5-point scale was used (0=poor, 1=fair, 2=good, 3=very good, 4=excellent).
Time Frame: Day 10
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Bisolviral
Number analyzed (Participants) | 97 | 98
percentage of participants
  Excellent | 2.1 | 2.0
  Very good | 11.3 | 16.3
  Good | 36.1 | 33.7
  Fair | 33.0 | 28.6
  Poor | 17.5 | 19.4
Statistical Analysis 1: Comparison: Placebo vs Bisolviral; Test type: Superiority or Other; p = 0.6954, Regression, Logistic; Odds Ratio (OR) = 1.1069, 95% CI 2-sided [0.666 to 1.840] — A value greater than one favours bisolviral

ADVERSE EVENTS:
Time Frame: From first nasal spray administration until the application discontinuation date plus one day, up to 11 days
Arm/Group | Placebo | Bisolviral
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.